CLINICAL TRIAL: NCT06097065
Title: Research on Potential Biomarkers of Prediabetes and Diabetes Based on MALDI-TOF MS Platform.
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhujiangzx
Record Dates: First submitted 2023-10-09; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-02

CONDITIONS: Prediabetes; Diabetes Mellitus; Gestational Diabetes Mellitus; Proteomics
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus; Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non pregnant people with prediabetes or diabetes: Non pregnancy meeting the diagnosis of prediabetes or diabetes.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test
- Non pregnant people with normal glucose tolerance: Non pregnant population with normal Oral Glucose Tolerance Test results.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test
- pregnant people with gestational diabetes mellitus: Pregnant people who meet the diagnosis of gestational diabetes.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test
- pregnant people with normal glucose tolerance: Pregnant people with normal Oral Glucose Tolerance Test results.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — Grouping based on detected oral glucose tolerance test results without any other intervention.

SUMMARY:
Through the MALDI-TOF MS platform, explore the proteomics and peptidomics differences of fasting serum/plasma and urine between non pregnant people with normal glucose tolerance test and prediabetes /diabetes patients, pregnant people with normal glucose tolerance test and pregnant diabetes patients respectively; To explore the role of its proteomics and peptidomics differences in the diagnosis of prediabetes and diabetes, and to establish a new method of differential diagnosis by using the omics data and key characteristic peaks to find potential new diagnostic markers.

DETAILED DESCRIPTION:
Prediabetes is a stage of abnormal glucose metabolism between normal blood glucose level and diabetes, which is a "gray zone" between normal and abnormal, including impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or both. It is a very important high-risk group of diabetes. Diabetes is a group of metabolic diseases characterized by hyperglycemia caused by a variety of causes. Gestational diabetes mellitus refers to varying degrees of abnormal glucose metabolism that occur during pregnancy. This project aims to detect differential feature peaks through MALDI-TOF MS technology between non pregnant people with normal glucose tolerance test and prediabetes/diabetes patients, pregnant people with normal glucose tolerance test and pregnant diabetes patients respectively and to establish a clinical predictive diagnostic model based on differences, and to evaluate the model.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for cases:

   Non pregnant people: the remaining fasting serum/plasma and urine samples of prediabetes/diabetes patients (prediabetes: IFG: FPG 6.1-6.9mmol/L, Blood glucose 2h after meal<7.8mmol/L（WHO）; IGT: FPG<7.0mmol/L, Blood glucose 2h after meal 7.8-11.1mmol/L（WHO）; diabetes: Typical symptoms of diabetes, FPG >= 7.0mmol/L or 75g OGTT 2h blood glucose >= 11.1mmol/L).

   Pregnant people: the remaining fasting serum/plasma and urine samples of gestational diabetes patients (75g OGTT test FPG >= 5.1mmol/L or 1h blood glucose >= 10.0mmol/L or 2h blood glucose >= 8.5mmol/L（IADPSG; ADA)).
2. Inclusion criteria of the controls were as follows:

Non pregnant people: the remaining fasting serum/plasma and urine samples of normal population for glucose tolerance test (FPG 3.9-6.1mmol/L,75g OGTT test 1h blood glucose 6.7-11.1mmol/L,75g OGTT test 2h blood glucose 3.6-7.8mmol/L).

Pregnant people: the remaining fasting serum/plasma and urine samples of people who do not meet the diagnostic criteria for gestational diabetes (3.9<=75g OGTT test FPG<5.1mmol/L,6.7 <= 1h blood glucose<10.0mmol/L,3.6<=2h blood glucose<8.5mmol/L).

-

Exclusion Criteria:

Common exclusion criteria for cases and control were as follows: The sample volume of serum/plasma/urine is less than 300ul; Improper storage of samples or repeated freezing and thawing; The serum /plasma has obvious hemolysis, lipemia or jaundice.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: (1) cases: Non pregnant people: the remaining fasting serum/plasma and urine samples of prediabetes/diabetes patients; Pregnant people: the remaining fasting serum/plasma and urine samples of gestational diabetes patients. (2) controls: (Non)pregnant people: the remaining fasting serum/plasma and urine samples of normal population.
Sampling Method: Non-Probability Sample
Enrollment: 2860 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and types of proteins/peptides differential characteristic peaks | one year
  Obtain the number and types of proteins/peptides differential characteristic peaks between the case group and the control group through data analysis.

SECONDARY OUTCOMES:
ROC curve and area under curve AUC of clinical predictive diagnostic model | one year
  Construct a clinical predictive diagnostic model based on the obtained proteins/peptides differential feature peaks and calculate the area under the ROC curve AUC to evaluate the predictive effect of the model.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Professor, Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China